CLINICAL TRIAL: NCT03311711
Title: Preparation for End-of-Life Decision Making in Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mi-Kyung Song, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099738; 1R01AG057714 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Dementia
Keywords: Alzheimer's Disease; Aging; Behavioral Research
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPIRIT-in person (Experimental): Patients and surrogates who participate in the SPIRIT intervention in person.
  Interventions: Behavioral: SPIRIT-in person
- SPIRIT-remote (Experimental): Patients and surrogates who participate in the SPIRIT intervention remotely, via teleconference.
  Interventions: Behavioral: SPIRIT-remote
- Usual care (Active Comparator): Patients and surrogates who receive the standard information about advance directives that is provided at the time of diagnosis.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: SPIRIT-in person — The SPIRIT-in person intervention adapted for dementia will include one session and will be conducted in a private room at the clinic. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention is expected to last 45-60 minutes.
  Arms: SPIRIT-in person
Behavioral: SPIRIT-remote — The SPIRIT-remote intervention adapted for dementia will include one session and will be conducted through teleconference. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention is expected to last 45-60 minutes.
  Arms: SPIRIT-remote
Behavioral: Usual care — Participants will receive the usual care that is provided through the clinic they receive care through. This may include completing advanced directives, referral to a support group, or referral to a social worker for further discussion about end of life issues.
  Other Names: Clinic standard of care
  Arms: Usual care

SUMMARY:
The proposed study will adapt and pilot test an efficacious advance care planning interventions, Sharing Patient's Illness Representations to Increase Trust (SPIRIT), with patients with mild dementia and their surrogates to promote open, honest discussions while such discussions about end-of-life care are possible. Patient and surrogate decision maker dyads will participate in a single SPIRIT session and will then have a follow up phone call 2-3 days later. One year after the SPIRIT session some surrogates will be contacted to provide additional feedback about the intervention.

DETAILED DESCRIPTION:
Progressive memory loss and impairment of reasoning and judgment are the main symptoms of dementia (including Alzheimer's Disease). For this reason, people in the early stages of dementia are encouraged to engage in advance care planning (ACP) while they are still competent to appoint a surrogate decision maker and meaningfully participate in ACP discussions with the surrogate.

The most common type of ACP is completing a medical power of attorney or living will, which does not require the patient and/or the family to understand the complexity of the medical decision-making process faced by the surrogate as the patient progresses to advanced disease. The failure to engage in ACP before the window of opportunity closes (i.e., before loss of decision making capacity) has serious adverse consequences with the greatest impact on the surrogate. As a matter of course in dementia, family members are left to make decisions regarding care transition, tube feeding, and other life-sustaining treatment without input from the patient and in the absence of a full understanding of the wishes, values and preferences of the patient.

To make an impact on the state of ACP for patients with dementia and their surrogates, the researchers will adapt and pilot test an efficacious ACP intervention, Sharing Patient's Illness Representations to Increase Trust (SPIRIT), with patients with mild dementia and their surrogates to promote open, honest discussions while such discussions about end-of-life care are possible. SPIRIT is a brief, scalable patient- and family-centered ACP intervention based on the Representational Approach to Patient Education with a goal to promote cognitive and emotional preparation for end-of-life decision making for patients with a serious or life-threatening illness and their surrogates. SPIRIT focuses on having both the patient and the surrogate fully understand end-of-life decision making in anticipation of a loss of decision-making capacity.

A panel of seven experts will provide feedback on adapting SPIRIT to persons with dementia and their surrogates, followed by pilot testing among the target population to refine the intervention. SPIRIT will also be adapted to a video conference format so that patients and surrogates can receive the intervention in their home. In this study, the SPIRIT intervention will be examined with a randomized clinical trial with three groups: SPIRIT-in person, SPIRIT-remote, and usual care. The researchers will recruit 120 dyads of patients with mild dementia and their surrogates, and the groups will be stratified by race (white vs non-white). The primary outcomes are patient and surrogate self-reported preparedness for end-of-life decision making which will be measured at baseline and shortly after the intervention (by phone in the next 2-3 days). Additionally, the researchers will compare the completion rates of advance directives among the three groups and the impact of the three treatment conditions perceived by surrogates at 1-year post intervention.

As of July 2020, recruitment of participants into the SPIRIT-in person study arm ceased in consideration of social distancing guidelines due to the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic. Participants enrolled after this date will be randomized to either the SPIRIT-remote or usual care study arms.

ELIGIBILITY:
Inclusion Criteria for Patients with Mild to Moderate Dementia:

* A diagnosis of mild to moderate dementia based on a Montreal Cognitive Assessment (MoCA) score greater than or equal to 13, or Mini-Mental State Examination (MMSE) score greater than or equal to 18
* Have access to a computer and internet connectivity in a private setting (either the patient or the surrogate has access to a computer and internet connectivity)
* Have decision-making capacity to consent to a low-risk study determined by a score greater than or equal to 11 on the University of California San Diego Brief Assessment of Capacity to Consent (UBACC)
* Able to understand and speak English

Exclusion Criteria for Patients with Mild to Moderate dementia:

* Lack of an available surrogate
* Uncompensated hearing deficits
* Speech impairment

Inclusion Criteria for Surrogates:

* 18 years or older (to serve as a surrogate decision-maker, the individual must be an adult)
* Be chosen by the patient to serve as a surrogate decision-maker
* Have access to a computer and internet connectivity in a private setting (either the patient or the surrogate has access to a computer and internet connectivity)
* Able to understand and speak English

Exclusion Criteria for Surrogates:

* Inability to complete questionnaires due to physical or cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, PhD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Assisted Living Facilities in the Metro Atlanta Area, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory Clinic Geriatrics, Atlanta, Georgia
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song MK, Ward SE, Hepburn K, Paul S, Kim H, Shah RC, Morhardt DJ, Medders L, Lah JJ, Clevenger CC. Can Persons with Dementia Meaningfully Participate in Advance Care Planning Discussions? A Mixed-Methods Study of SPIRIT. J Palliat Med. 2019 Nov;22(11):1410-1416. doi: 10.1089/jpm.2019.0088. Epub 2019 Aug 2. PMID 31373868
- [Derived] Song MK, Ward SE, Hepburn K, Paul S, Shah RC, Morhardt DJ. SPIRIT advance care planning intervention in early stage dementias: An NIH stage I behavioral intervention development trial. Contemp Clin Trials. 2018 Aug;71:55-62. doi: 10.1016/j.cct.2018.06.005. Epub 2018 Jun 2. PMID 29870867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from healthcare clinics in Georgia and Illinois, USA. Participant enrollment began May 4, 2018. Follow-up for the 2-3 day post-intervention assessment was completed by February 3, 2022 and follow up for the 12 months post-intervention time point was completed by December 7, 2022.
Pre-assignment Details: In July 2020 the protocol was modified, eliminating the SPIRIT-in person intervention due to the coronavirus disease 2019 (COVID-19) pandemic which prohibited in person research visits. The study design changed to SPIRIT-remote versus usual care and a new randomization method was initiated for the two arm design. Due to the change in randomization method mid-study, participants enrolled before and after the randomization change are analyzed separately (as original or modified randomization).
Groups:
- SPIRIT-in Person - Persons With Dementia, Original Randomization: Persons with dementia participating in the SPIRIT intervention in person, during the original randomization design.
  SPIRIT-in person: The SPIRIT-in person intervention adapted for dementia includes one session and is conducted in a private room at the clinic. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- SPIRIT-in Person - Surrogates, Original Randomization: Surrogates participating in the SPIRIT intervention in person, during the original randomization design.
  SPIRIT-in person: The SPIRIT-in person intervention adapted for dementia includes one session and is conducted in a private room at the clinic. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- SPIRIT-remote - Persons With Dementia, Original Randomization: Persons with dementia participating in the SPIRIT intervention remotely, via teleconference, during the original randomization design.
  SPIRIT-remote: The SPIRIT-remote intervention adapted for dementia includes one session and is conducted through teleconference. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- SPIRIT-remote - Surrogates, Original Randomization: Surrogates participating in the SPIRIT intervention remotely, via teleconference, during the original randomization design.
  SPIRIT-remote: The SPIRIT-remote intervention adapted for dementia includes one session and is conducted through teleconference. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- Usual Care - Persons With Dementia, Original Randomization: Persons with dementia receiving the standard information about advance directives that is provided at the time of diagnosis, during the original randomization design.
  Usual care: Participants receive the usual care that is provided through the clinic they receive care through. This may include completing advanced directives, referral to a support group, or referral to a social worker for further discussion about end of life issues.
- Usual Care - Surrogates, Original Randomization: Surrogates receiving the standard information about advance directives that is provided at the time of diagnosis, during the original randomization design.
  Usual care: Participants receive the usual care that is provided through the clinic they receive care through. This may include completing advanced directives, referral to a support group, or referral to a social worker for further discussion about end of life issues.
- SPIRIT-remote - Persons With Dementia, Modified Randomization: Persons with dementia participating in the SPIRIT intervention remotely, via teleconference, during the modified randomization design.
  SPIRIT-remote: The SPIRIT-remote intervention adapted for dementia includes one session and is conducted through teleconference. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- SPIRIT-remote - Surrogates, Modified Randomization: Surrogates participating in the SPIRIT intervention remotely, via teleconference, during the modified randomization design.
  SPIRIT-remote: The SPIRIT-remote intervention adapted for dementia includes one session and is conducted through teleconference. SPIRIT is a structured psychoeducational intervention, targeting both patient and surrogate. The SPIRIT intervention assists patients in clarifying their end-of-life preferences and helps surrogates understand the patient's wishes and prepare for the surrogate role. The intervention lasts 45-60 minutes.
- Usual Care - Persons With Dementia, Modified Randomization: Persons with dementia receiving the standard information about advance directives that is provided at the time of diagnosis, during the modified randomization design.
  Usual care: Participants receive the usual care that is provided through the clinic they receive care through. This may include completing advanced directives, referral to a support group, or referral to a social worker for further discussion about end of life issues.
- Usual Care - Surrogates, Modified Randomization: Surrogates receiving the standard information about advance directives that is provided at the time of diagnosis, during the modified randomization design.
  Usual care: Participants receive the usual care that is provided through the clinic they receive care through. This may include completing advanced directives, referral to a support group, or referral to a social worker for further discussion about end of life issues.
Period: Overall Study
Arm/Group | SPIRIT-in Person - Persons With Dementia, Original Randomization | SPIRIT-in Person - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Original Randomization | SPIRIT-remote - Surrogates, Original Randomization | Usual Care - Persons With Dementia, Original Randomization | Usual Care - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Modified Randomization | SPIRIT-remote - Surrogates, Modified Randomization | Usual Care - Persons With Dementia, Modified Randomization | Usual Care - Surrogates, Modified Randomization
Started | 15 | 15 | 12 | 12 | 15 | 15 | 40 | 40 | 39 | 39
Completed | 11 | 11 | 12 | 12 | 15 | 15 | 35 | 35 | 38 | 38
Not Completed | 4 | 4 | 0 | 0 | 0 | 0 | 5 | 5 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death of dyad partner | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SPIRIT-in Person - Persons With Dementia, Original Randomization: Persons with dementia participating in the SPIRIT intervention in person, during the original randomization design.
- SPIRIT-in Person - Surrogates, Original Randomization: Surrogates participating in the SPIRIT intervention in person, during the original randomization design.
- SPIRIT-remote - Persons With Dementia, Original Randomization: Persons with dementia participating in the SPIRIT intervention remotely, via teleconference, during the original randomization design.
- SPIRIT-remote - Surrogates, Original Randomization: Surrogates participating in the SPIRIT intervention remotely, via teleconference, during the original randomization design.
- Usual Care - Persons With Dementia, Original Randomization: Persons with dementia receiving the standard information about advance directives that is provided at the time of diagnosis, during the original randomization design.
- Usual Care - Surrogates, Original Randomization: Surrogates receiving the standard information about advance directives that is provided at the time of diagnosis, during the original randomization design.
- SPIRIT-remote - Persons With Dementia, Modified Randomization: Persons with dementia participating in the SPIRIT intervention remotely, via teleconference, during the modified randomization design.
- SPIRIT-remote - Surrogates, Modified Randomization: Surrogates participating in the SPIRIT intervention remotely, via teleconference, during the modified randomization design.
- Usual Care - Persons With Dementia, Modified Randomization: Persons with dementia receiving the standard information about advance directives that is provided at the time of diagnosis, during the modified randomization design.
- Usual Care - Surrogates, Modified Randomization: Surrogates receiving the standard information about advance directives that is provided at the time of diagnosis, during the modified randomization design.
- Total: Total of all reporting groups
Arm/Group | SPIRIT-in Person - Persons With Dementia, Original Randomization | SPIRIT-in Person - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Original Randomization | SPIRIT-remote - Surrogates, Original Randomization | Usual Care - Persons With Dementia, Original Randomization | Usual Care - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Modified Randomization | SPIRIT-remote - Surrogates, Modified Randomization | Usual Care - Persons With Dementia, Modified Randomization | Usual Care - Surrogates, Modified Randomization | Total
Number analyzed (Participants) | 15 | 15 | 12 | 12 | 15 | 15 | 40 | 40 | 39 | 39 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.53 (10.66) | 65.20 (15.36) | 78.83 (8.25) | 67.58 (7.83) | 74.00 (9.00) | 62.20 (12.04) | 74.07 (8.50) | 65.60 (12.89) | 72.82 (8.09) | 68.85 (9.62) | 70.34 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 5 | 11 | 8 | 9 | 26 | 27 | 18 | 24 | 146
  Male | 6 | 6 | 7 | 1 | 7 | 6 | 14 | 13 | 21 | 15 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 6
  Not Hispanic or Latino | 15 | 15 | 12 | 12 | 15 | 15 | 39 | 39 | 37 | 37 | 236
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 5 | 5 | 5 | 3 | 3 | 8 | 7 | 5 | 6 | 52
  White | 10 | 10 | 7 | 7 | 11 | 12 | 32 | 32 | 32 | 32 | 185
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 12 | 12 | 15 | 15 | 40 | 40 | 39 | 39 | 242

OUTCOME MEASURES:

1. Primary Outcome: Dyad Congruence With Goals-of-Care Tool
Description: Dyad congruence was assessed using the Goals-of-Care Tool which has been modified to include two scenarios relevant to the context of dementia. There are three response options: "The goals of care should focus on delaying my death no matter what, and thus I want to continue life-sustaining treatment", "The goals of care should focus on my comfort and peace, and thus I do not want life-sustaining treatment", and "I am not sure". Persons with dementia and surrogates complete this tool independently and their responses are then compared to determine dyad congruence (either congruent in both scenarios or incongruent). If both members of the dyad endorse "I am not sure", they are considered incongruent.
Time Frame: Baseline, follow up phone call at 2-3 days post-intervention
Population: The number of participants analyzed reflects the number of person with dementia and surrogate dyads (two persons per dyad). This analysis includes dyads who completed the indicated study visit. Three dyads from the SPIRIT-in person original randomization, and 3 dyads from the SPIRIT-remote modified randomization did not complete the 2-3 day post-intervention follow up visit.
Measure: Count of Participants; unit: Participants
Groups:
- SPIRIT-in Person, Original Randomization: Person with dementia and surrogate dyads participating in the SPIRIT intervention in person, during the original randomization design.
- SPIRIT-remote, Original Randomization: Person with dementia and surrogate dyads participating in the SPIRIT remotely, during the original randomization design.
- Usual Care, Original Randomization: Person with dementia and surrogate dyads receiving usual care, during the original randomization design.
- SPIRIT-remote, Modified Randomization: Person with dementia and surrogate dyads participating in the SPIRIT remotely, during the modified randomization design.
- Usual Care, Modified Randomization: Person with dementia and surrogate dyads receiving usual care, during the modified randomization design.
Arm/Group | SPIRIT-in Person, Original Randomization | SPIRIT-remote, Original Randomization | Usual Care, Original Randomization | SPIRIT-remote, Modified Randomization | Usual Care, Modified Randomization
Number analyzed (Participants) | 15 | 12 | 15 | 40 | 39
Participants
  Number of Congruent Dyads at Baseline | 9 | 4 | 11 | 24 | 30
  Number of Incongruent Dyads at Baseline | 6 | 8 | 4 | 16 | 9
  Number of Congruent Dyads at 2-3 Days Post-intervention: number analyzed (Participants) | 12 | 12 | 15 | 37 | 39
  Number of Congruent Dyads at 2-3 Days Post-intervention | 11 | 9 | 11 | 34 | 32
  Number of Incongruent Dyads at 2-3 Days Post-intervention: number analyzed (Participants) | 12 | 12 | 15 | 37 | 39
  Number of Incongruent Dyads at 2-3 Days Post-intervention | 1 | 3 | 4 | 3 | 7

2. Primary Outcome: Surrogate's Decision Making Confidence (DMC) Scale Score Among Phase II Participants
Description: Surrogate decision-making confidence is measured using the 5-item Decision Making Confidence (DMC) scale. DMC assesses a surrogate's confidence in knowing the patient's wishes, ability to make treatment decisions even in a highly stressful situation, ability to seek information about risks and benefits of medical choices, ability to handle unwanted pressure from others, and ability to communicate with providers about the patient's wishes. Surrogates indicate how confident they are about making medical decisions, if the patient becomes unable to make their own decisions, by their level of agreement with statements along a scale of (0) "not confident at all" to (4) "Very confident". Total scores range from 0 - 20, with higher scores indicating greater confidence.
Time Frame: Baseline, follow up phone call at 2-3 days post-intervention
Population: This analysis includes participants who completed the indicated study visit. Three dyads from the SPIRIT-in person original randomization, and 3 dyads from the SPIRIT-remote modified randomization did not complete the 2-3 day post-intervention follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT-in Person - Surrogates, Original Randomization | SPIRIT-remote - Surrogates, Original Randomization | Usual Care - Surrogates, Original Randomization | SPIRIT-remote - Surrogates, Modified Randomization | Usual Care - Surrogates, Modified Randomization
Number analyzed (Participants) | 15 | 12 | 15 | 40 | 39
score on a scale
  Baseline | 18.40 (1.24) | 18.08 (1.73) | 18.20 (1.78) | 18.33 (2.21) | 18.10 (2.10)
  2-3 Days Post-intervention: number analyzed (Participants) | 12 | 12 | 15 | 37 | 39
  2-3 Days Post-intervention | 19.08 (1.24) | 18.42 (1.83) | 19.07 (1.39) | 19.35 (1.14) | 19.05 (1.23)

3. Primary Outcome: Surrogate's Overall Preparedness Scale
Description: The Overall Preparedness Scale for end-of-life decision making for surrogates is a 23-item investigator-developed measure. The measure assesses the level of preparedness for end-of-life decision making in the cognitive, emotional, and behavioral dimensions on a 4-point scale (1=strongly disagree to 4=strongly agree). Total scores range from 23 to 92, with higher scores indicating higher levels of preparedness.
Time Frame: Baseline, follow up phone call at 2-3 days post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT-in Person - Surrogates, Original Randomization | SPIRIT-remote - Surrogates, Original Randomization | Usual Care - Surrogates, Original Randomization | SPIRIT-remote - Surrogates, Modified Randomization | Usual Care - Surrogates, Modified Randomization
Number analyzed (Participants) | 15 | 12 | 15 | 40 | 39
score on a scale
  Baseline | 75.27 (6.91) | 75.75 (9.76) | 75.53 (9.15) | 72.15 (8.82) | 74.69 (7.42)
  2-3 Days Post-intervention: number analyzed (Participants) | 12 | 12 | 15 | 37 | 39
  2-3 Days Post-intervention | 83.75 (4.05) | 76.92 (8.18) | 78.73 (8.42) | 81.50 (6.97) | 77.80 (8.32)

4. Secondary Outcome: Completion of Advance Directives Among Phase II Participants
Description: At the Baseline visit, participants were asked if they had already completed an advance directive. Medical records were reviewed to determine if the patient completed an advance directive (a medical power of attorney or living will) by 12 months post-intervention. If there was no documentation in the medical record, the surrogate was contacted to get confirmation on the status of the Advance Directive.
Time Frame: Baseline, up to 12 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SPIRIT-in Person - Persons With Dementia, Original Randomization | SPIRIT-remote - Persons With Dementia, Original Randomization | Usual Care - Persons With Dementia, Original Randomization | SPIRIT-remote - Persons With Dementia, Modified Randomization | Usual Care - Persons With Dementia, Modified Randomization
Number analyzed (Participants) | 15 | 12 | 15 | 40 | 39
Participants
  Baseline - Complete | 10 | 9 | 14 | 33 | 30
  Baseline - Incomplete | 5 | 3 | 1 | 7 | 9
  12-month cumulative - Complete | 12 | 12 | 15 | 38 | 38
  12-month cumulative - Incomplete | 3 | 0 | 0 | 2 | 1

5. Secondary Outcome: Patient's Overall Preparedness Scale
Description: The Overall Preparedness Scale for end-of-life decision making for patients is a 22 item investigator-developed measure. The measure assesses the level of preparedness for end-of-life decision making in the cognitive, emotional, and behavioral dimensions on a 4-point scale (1=strongly disagree to 4=strongly agree). Total scores range from 22 to 88, with higher scores indicating higher levels of preparedness.
Time Frame: Baseline, follow up phone call at 2-3 days post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT-in Person - Persons With Dementia, Original Randomization | SPIRIT-remote - Persons With Dementia, Original Randomization | Usual Care - Persons With Dementia, Original Randomization | SPIRIT-remote - Persons With Dementia, Modified Randomization | Usual Care - Persons With Dementia, Modified Randomization
Number analyzed (Participants) | 15 | 12 | 15 | 40 | 39
score on a scale
  Baseline | 55.40 (6.97) | 54.67 (5.14) | 54.07 (7.54) | 54.90 (5.71) | 53.50 (5.96)
  2-3 Days Post-intervention: number analyzed (Participants) | 12 | 12 | 15 | 37 | 39
  2-3 Days Post-intervention | 57.83 (6.60) | 58.57 (5.31) | 54.93 (9.03) | 58.78 (5.20) | 54.69 (5.50)

ADVERSE EVENTS:
Time Frame: Adverse events were documented during the intervention session (Day 1). Known deaths that occurred up to the 12 month assessment were documented.
Description: Only adverse events related to the intervention, such as emotional distress, were documented during the intervention session. Due to the population being examined and the nature of this study, deaths are not considered as an adverse event in this population, however, known deaths occurring up to the 12 month assessment were documented.
Arm/Group | SPIRIT-in Person - Persons With Dementia, Original Randomization | SPIRIT-in Person - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Original Randomization | SPIRIT-remote - Surrogates, Original Randomization | Usual Care - Persons With Dementia, Original Randomization | Usual Care - Surrogates, Original Randomization | SPIRIT-remote - Persons With Dementia, Modified Randomization | SPIRIT-remote - Surrogates, Modified Randomization | Usual Care - Persons With Dementia, Modified Randomization | Usual Care - Surrogates, Modified Randomization
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/15 | 0/12 | 0/12 | 0/15 | 0/15 | 1/40 | 0/40 | 1/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12 | 0/12 | 0/15 | 0/15 | 0/40 | 0/40 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12 | 0/12 | 0/15 | 0/15 | 0/40 | 0/40 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03311711/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03311711/ICF_000.pdf